CLINICAL TRIAL: NCT06706440
Title: The Study of the Natural Way of Development of External Pancreatic Fistulas in Children with Necrotizing Pancreatitis
Status: Completed | Type: Observational
Sponsor: Moscow Regional Research and Clinical Institute (MONIKI) (Other Government)
Responsible Party: Sponsor
Other Study IDs: 16/05.11.2024
Record Dates: First submitted 2024-11-20; First posted 2024-11-26 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Children; Pancreatic Fistula; Pancreatitis,Acute Necrotizing; Pancreatitis, Acute
Keywords: Children; Acute necrotizing pancreatitis; Pancreatic fistula
MeSH Terms: conditions — Pancreatic Fistula; Pancreatitis, Acute Necrotizing; Pancreatitis | interventions — Observation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- children with external pancreatic fistula: children who have suffered acute necrotizing pacreatitis and undergone drainage of parapancreatic accumulations, with the development of an external pancreatic fistula
  Interventions: Other: no intervention, observational study

INTERVENTIONS:
Other: no intervention, observational study — Only data will be taken of patient's file.

SUMMARY:
The external pancreatic fistula (EPF) is characterized by the leakage of pancreatic juice outward through an area of skinor through a drainage tube.

The leakage of pancreatic juice occurs due to the rupture of the pancreatic duct (PD) caused by the destruction of pancreatic tissue. EPF can cause deterioration in the patient's condition due to the leakage of protein-rich pancreatic juice outward, as well as the increased risk of skin irritation and infection.

DETAILED DESCRIPTION:
The treatment of EPF has traditionally been conservative, including the nutritional support in an attempt to reduce pancreatic secretion, or total parenteral nutrition with antisecretory therapy (octreotide). In cases where the conservative therapy has proved to be ineffective, there has been performed the surgical treatment. The cases of successful treatment of EPF by endoscopic transpapillary drainage have been reported in the literature as an effective and minimally invasive therapeutic alternative to the surgery for the treatment of EPF. However, the endoscopic transpapillary drainage is usually ineffective in patients with the complete PD failure. The complete PD failure in the presence of the functional pancreas above the failure results in the disconnected pancreatic duct syndrome.

Sepsis, infection, electrolyte disturbances, malnutrition, and infections are commonly seen in patients with high-output EPF. In addition, there has occasionally been reported the spontaneous closure of low-output EPF. However, there are no data on the natural history of EPF.

The aim of this study is to evaluate the natural clinical history of EPF in children with necrotizing pancreatitis by examining the outcomes and the complications of the conservative treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patient or legal representative consent
* External pancreatic fistula
* Age from 0-18 years
* Moderate severe (MSAP) or severe acute pancreatitis (SAP) according to Atlanta criteria revisited in 2012
* Acute Pancreatitis was defined in case of the presence of at least two of the three criteria according to the classification developed by the INSPPIRE (International Study Group of Pediatric Pancreatitis: In Search for a Cure) group: abdominal pain consistent with the diagnostic hypothesis; serum amylase and/or lipase increased by ≥3 times; imaging results typical of AP: abdominal ultrasound and/or contrast-enhanced CT.

Exclusion Criteria:

* Mild acute pancreatitis
* Chronic pancreatitis
* No consent from patient or legal representative

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Moscow Regional Scientific Research Clinical Institute named after M.F. Vladimirsky
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2024-11-11 (Actual); Primary Completion 2025-01-10 (Actual); Study Completion 2025-02-18 (Actual)

PRIMARY OUTCOMES:
The duration of pancreatic fistula functioning | From the day of surgery to the end of treatment (9 months)
  based on testing serum lipase and/or amylase concentrations in drained fluid, imaging results: ultrasound (US), spiral computed tomography (SCT), magnetic resonance imaging (MRI), fistolography

SECONDARY OUTCOMES:
The level of damage to the main pancreatic duct | From the day of surgery to the end of treatment (9 months)
  MRCP
The duration of hospital stay | From the day of surgery to the end of treatment (9 months)
The mortality | From enrollment to the end of treatment (9 month)
The dynamics of the total protein | From enrollment to the end of treatment (9 month)
  total protein (G/L)
The effect of the etiologic factor on the duration of the external pancreatic fistula functioning | From enrollment to the end of treatment (9 month)
  number of days of functioning of the external pancreatic fistula depending on the etiological factor: trauma, ERCP, common bile duct stone, idiopathic, hypertriglyceridemia, alcohol
The dynamics of the drain tube fluid amylase | From enrollment to the end of treatment (9 month)
  drain tube fluid amylase (U/L)
The dynamics of the blood amylase | From enrollment to the end of treatment (9 month)
  blood amylase (U/L)

CONTACTS AND LOCATIONS:
Overall Officials: Dmitriy А Pyhteev, PhD, Study Director — Head of the Department of Pediatric Surgery; Leonid M Elin, Principal Investigator — Moscow Regional Scientific Research Clinical Institute named after M.F. Vladimirsky
Locations (1):
- Moscow Regional Scientific Research Clinical Institute named after M.F. Vladimirsky, Moscow, Russia

IPD SHARING:
Plan to Share IPD: Yes
A complete dataset can be provided upon reasoned request